CLINICAL TRIAL: NCT00601328
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalency Study of Calcitriol Tablets, 0.25 mg, Under Fasting Conditions
Brief Title: Bioequivalency Study of Calcitriol Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth A. Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CALC-07
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Secondary Hyperparathyroidism; Hypocalcemia
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypocalcemia | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Calcitriol

SUMMARY:
The objective of this study was to assess the bioequivalence of Roxane Laboratories' Calcitriol capsules, 0.25 mcg, to ROCALTROL® capsules, 0.25 mcg (Roche) using a single-dose, 2-treatment, 2-period, crossover design, under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Calcitriol or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2003-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Fourteen day washout

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Morrison, DO, Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri, United States